CLINICAL TRIAL: NCT00509938
Title: Safety and Efficacy of Human Lactoferrin hLF1-11 for the Treatment of Infectious Complications Among Haematopoietic Stem Cell Transplant Recipients Part A: Clinical Study Protocol SC12: Safety of a Single Dose of 5 mg of hLF1-11 Given to Autologous Haematopoietic Stem Cell Transplant Recipients
Brief Title: Safety of a Single Dose of 5 mg of hLF1-11 Given to Autologous Haematopoietic Stem Cell Transplant Recipients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AM-Pharma (Industry)
Responsible Party: Jacques Arend MD, VP Medical Development, AM-Pharma
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AMP 02-01; SC12; IS 044096
Record Dates: First submitted 2007-07-31; First posted 2007-08-01 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Hematopoietic Stem Cell Transplantation; Bacterial Infections and Mycoses
Keywords: immunocompromized; hLF1-11; antimicrobial; peptide; lactoferrin
MeSH Terms: conditions — Bacterial Infections and Mycoses | interventions — lactoferrin (1-11), human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): 5mg hLF1-11, single dose iv
  Interventions: Drug: human lactoferrin peptide 1-11

INTERVENTIONS:
Drug: human lactoferrin peptide 1-11 — Each subject will receive a single intravenous dose of hLF1-11 given in a volume of 20mL given over 20 minutes i.e. 1mL/per minute.

SUMMARY:
The safety and tolerability of hLF 1-11 has to be established first in HSCT recipients who are at risk of developing, but have not yet developed, infectious complications due to invasive fungal disease. These patients are different from healthy volunteers because they have received myeloablative treatment which not only arrests haematopoiesis resulting in neutropenia but also induces mucosal barrier injury both of which predispose to infections which typically occur during the week after transplant. It is therefore essential to know that hLF 1-11 is when given during neutropenia and mucosal barrier injury before infections ensue

DETAILED DESCRIPTION:
Background:

Human lactoferrin (hLF) is a glycoprotein containing 692 amino acids and found in the saliva, milk, tears, and other body fluids. Peptide representing the first cationic domain, i.e. a peptide comprising the first eleven residues of hLF (further referred to as hLF1-11) was significantly more effective than the full length hLF or the peptide representing the second cationic domain in killing a variety of bacteria in vivo. The mechanism of action comprises a number of independent factors. The classical way to explain the efficacy is the direct killing effect, which typically is observed in vitro at relatively high concentrations. The results of in vitro and in vivo experiments suggest that the mechanism of action is predominantly through the intermediary of cells and/or components of the host as opposed to a direct interaction with the pathogen.

The objective is to develop hLF1-11 as an effective and safe antibacterial and antifungal for the treatment of fungal and bacterial infections that develop during the neutropenia that results from myeloablative therapy to prepare for a haematopoietic stem cell transplant (HSCT) formerly referred to as bone marrow transplant. Rates of infection and related morbidity are high in this population making it an attractive target for testing clinically the proof-of-principle that hLF1-11 can provided effective treatment. Subsequently, hLF1-11 will be developed further as a systemic antifungal agent.

ELIGIBILITY:
Inclusion Criteria:

* admitted for an autologous HSCT after myeloablative therapy with high-dose melfalan
* managed with a 4-lumen central venous catheter
* BMI <30
* able and willing to participate
* has provided written informed consent
* there is no medical reason for exclusion
* has adequate renal function (creatinine <110 µmol/L (man); <90 µmol/L (woman))
* has adequate liver function (ASAT <40 U; ALAT <45 U; bilirubin <10µmol/L)
* has no known allergy to lactoferrin
* has no history of hepatitis and is not HIV seropositive
* if a woman, functionally post-menopausal

Exclusion Criteria:

* A history of, or presence of, significant respiratory, cardiovascular, neurological, haematological, endocrine, gastrointestinal, hepatic or renal disease or other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs (as judged clinically relevant by the investigator).
* Participation in a study with a new chemical entity or new molecular entity 3 months before or participation in a study with a registered drug less than 5 times of the half life of the registered drug before entering the study.
* A clinically relevant history of intolerance or hypersensitivity to the study drug, or its additives and excipients in the intravenous formulation.
* Evidence of having serum hepatitis or carrying the hepatitis B surface antigen or Hepatitis C antibodies or being HIV positive.
* Subjects, who in the opinion of the investigator should not, for reasons of safety, participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-03; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability by recording the vital signs, clinical chemistry, local tolerability and adverse events during the study | 28 Days

SECONDARY OUTCOMES:
formation of antibodies anti-hLF 1-11 during the study. | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: J.P. Donnelly, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- UMC St. Radboud, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Velden WJ, van Iersel TM, Blijlevens NM, Donnelly JP. Safety and tolerability of the antimicrobial peptide human lactoferrin 1-11 (hLF1-11). BMC Med. 2009 Sep 8;7:44. doi: 10.1186/1741-7015-7-44. PMID 19735580